CLINICAL TRIAL: NCT04422977
Title: Serological Study of the Exposure of Personnel to Sars-cov-2 in an Urban Hospital Two Months After Managing an Influx of COVID Patients 19
Brief Title: Serological Study of the Exposure of Personnel to COVID-19
Acronym: SEROPHUGAC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Saint Joseph Saint Luc de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: SEROPHUGAC
Record Dates: First submitted 2020-06-05; First posted 2020-06-09 (Actual); Last update posted 2024-04-04 (Actual); Status verified 2024-04

CONDITIONS: Sars-CoV2

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CoVID exposure (Other)
  Interventions: Diagnostic Test: Sars-Cov-2 serology

INTERVENTIONS:
Diagnostic Test: Sars-Cov-2 serology — Measurement of overall seroprevalence of SARS-Cov-2 in an hospital staff
  Other Names: serology

SUMMARY:
A seroconversion test for SARS-Cov-2 will be offered to all the employees of a care institution, which has treated 240 patients hospitalized for COVID disease between 28/02 and 30/04/2020. The seroconversion test will be with a questionnaire to determine:

* whether the subject has shown signs of infection in the last 3 recent months
* if the subject has been in contact with COVID-diagnosed subjects (RT-PCR diagnosis or scanner) outside of the activity or within the professional activity (patient or colleague)
* Working conditions during the period
* The level of knowledge and respect of the barrier measures practices.
* Respect for distance during meals professional. Overall seroprevalence and stratified seroprevalence by care and administrative areas will be determined.

ELIGIBILITY:
Inclusion Criteria:

* Subject who worked at Saint Joseph Saint Luke's Hospital during the epidemic wave (male or female).

  * Free and informed consent
  * Social security affiliation

Exclusion Criteria:

* Subject refusal
* Subject on leave during the entire period

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 957 (Actual)
Dates: Start 2020-06-08 (Actual); Primary Completion 2020-07-10 (Actual); Study Completion 2020-07-10 (Actual)

PRIMARY OUTCOMES:
Measurement of overall seroprevalence of SARS-Cov-2 in an hospital staff with a seroconversion test for SARS-Cov-2 | 1 month
  Measurement of overall seroprevalence of SARS-Cov-2 in an hospital staff

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier St Joseph St Luc, Lyon, France

REFERENCES:
- [Derived] Vivier E, Pariset C, Rio S, Armand S, Doroszewski F, Richard D, Chardon M, Romero G, Metral P, Pecquet M, Didelot A. Specific exposure of ICU staff to SARS-CoV-2 seropositivity: a wide seroprevalence study in a French city-center hospital. Ann Intensive Care. 2021 May 13;11(1):75. doi: 10.1186/s13613-021-00868-8. PMID 33987718